CLINICAL TRIAL: NCT02116517
Title: Phase 3 Study; Effects of Green Tea Extract on Obese Women With High Level of Low Density Lipoprotein (LDL): a Randomized, Double-blinded, and Cross-over Placebo-controlled Clinical Trial
Brief Title: Effects of Green Tea Extract on Obese Women With High Level of LDL
Acronym: GTE-LDL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Dr, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 100WFA2200449
Record Dates: First submitted 2014-04-04; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2013-12

CONDITIONS: Obese; Hyperlipidemia
Keywords: obese women; high LDL-C
MeSH Terms: conditions — Obesity; Hyperlipidemias | interventions — Tea; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- green tea extract first (Experimental): green tea extract (EGCG) 500mg tid for 6 weeks, then wash-out for 2 weeks, and finally cellulose 500mg tid for 6 weeks total 14 weeks
  Interventions: Dietary Supplement: green tea extract; Dietary Supplement: Placebo
- Placebo first (Placebo Comparator): cellulose 500mg tid for 6 weeks, then wash-out for 2 weeks, and finally EGCG 500mg tid for 6 weeks total 14 weeks
  Interventions: Dietary Supplement: green tea extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: green tea extract — 500 mg three times per day
  Other Names: EGCG
Dietary Supplement: Placebo — cellulose 500mg three times a day for 6 weeks
  Other Names: cellulose

SUMMARY:
Green tea is one of the most popular beverages in the world. It is believed to have beneficial effect in prevention and treatment of many diseases, one of which is reducing LDL-C. The aim of the study is to examine the effect of supplement containing GTE on obese with high LDL level.

DETAILED DESCRIPTION:
Randomized, double-blind, crossover placebo-controlled clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years
2. body mass index (BMI) >= 27 kg/m2
3. fasting low-density-lipoprotein cholesterol (LDL) >= 130mg/dl and (4) willing to participate in this trial.

Exclusion Criteria:

1. serum alanine transaminase > 80 U/L
2. serum creatinine > 1.8 mg/dl
3. breast feeding or pregnancy
4. heart failure, acute myocardial infarction, stroke, heavy injury
5. any other conditions not suitable for trial as evaluated by the physician. -

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
percentage of reduction of LDL-C | 6 weeks of treatment
  level of LDL-C before intervention minus level of LDL-C after intervention equal to reduction of LDL-C, percentage of reduction of LDL-C equal to the level of reduction of LDL-C divided by level of LDL-C before intervention

SECONDARY OUTCOMES:
HDL-C | 6 weeks
  serum level of high density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, PhD, MD, Study Chair — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Liu CY, Huang CJ, Huang LH, Chen IJ, Chiu JP, Hsu CH. Effects of green tea extract on insulin resistance and glucagon-like peptide 1 in patients with type 2 diabetes and lipid abnormalities: a randomized, double-blinded, and placebo-controlled trial. PLoS One. 2014 Mar 10;9(3):e91163. doi: 10.1371/journal.pone.0091163. eCollection 2014. PMID 24614112
- [Background] Hsu CH, Liao YL, Lin SC, Tsai TH, Huang CJ, Chou P. Does supplementation with green tea extract improve insulin resistance in obese type 2 diabetics? A randomized, double-blind, and placebo-controlled clinical trial. Altern Med Rev. 2011 Jun;16(2):157-63. PMID 21649457
- [Background] Hsu CH, Tsai TH, Kao YH, Hwang KC, Tseng TY, Chou P. Effect of green tea extract on obese women: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2008 Jun;27(3):363-70. doi: 10.1016/j.clnu.2008.03.007. Epub 2008 May 12. PMID 18468736
- [Derived] Huang LH, Liu CY, Wang LY, Huang CJ, Hsu CH. Effects of green tea extract on overweight and obese women with high levels of low density-lipoprotein-cholesterol (LDL-C): a randomised, double-blind, and cross-over placebo-controlled clinical trial. BMC Complement Altern Med. 2018 Nov 6;18(1):294. doi: 10.1186/s12906-018-2355-x. PMID 30400924